CLINICAL TRIAL: NCT00996034
Title: 123I-5-IA SPECT Imaging of Nicotinic Receptors and Effects of Nicotine Vaccine
Brief Title: Nicotine Vaccination and Nicotinic Receptor Occupancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Nabi Biopharmaceuticals (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0804003655; R21DA024388 (NIH)
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Nicotine Dependence
Keywords: Nicotine, SPECT, vaccine, receptor
MeSH Terms: conditions — Tobacco Use Disorder | interventions — NicVAX; 5-iodo-3-(2-azetidinylmethoxy)pyridine; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy Smoker (Experimental): There is only one arm to the study. All subjects will receive NicVax, [123I]5-I-A-85380,and Nicotine bitartrate.
  Interventions: Biological: NicVAX; Radiation: [123I]5-IA-85380; Drug: Nicotine bitartrate

INTERVENTIONS:
Biological: NicVAX — 1.0 mL of Nicotine Conjugate Vaccine(x4), I.M. at 3 week intervals between SPECT studies
  Other Names: Nicotine Conjugate Vaccine
Radiation: [123I]5-IA-85380 — up to 10 mCi of [123I]5-IA-85380, I.V. on each of two SPECT Scan days
  Other Names: 5-IA
Drug: Nicotine bitartrate — 0.5-1.5 mg of Nicotine bitartrate, I.V. on each of two SPECT Scan days
  Other Names: IV nicotine

SUMMARY:
This is a molecular imaging research study designed to examine how much nicotine gets into the brain before and after vaccination with NicVAX, a nicotine vaccine developed by Nabi Biopharmaceuticals. NicVAX (Nicotine Conjugate Vaccine) is an investigational vaccine designed as an aid to smoking cessation and long-term abstinence, as well as an aid to prevent relapses of a treated smoker.

In this project we want to understand the degree to which NicVAX administration changes how much nicotine enters the brain in smokers.

DETAILED DESCRIPTION:
The purpose of the present study is to examine the occupancy of brain β2-containing nicotinic acetylcholine receptors (β2-nAChR) by nicotine both at baseline and following administration of a nicotine vaccine. The number of brain β2-nAChR and the amount of nicotine occupancy both before and after vaccination will be measured using the nicotinic agonist [123I]5-IA-85380 ([123I]5-IA) and single photon emission computed tomography (SPECT). [123I]5-IA will be administered using the bolus plus constant infusion paradigm to smokers abstinent for 4-9 days (time period necessary for nicotine and pharmacological active metabolites to clear from brain). Three baseline SPECT images will be obtained after equilibrium has been reached (~6 hours into the [123I]5-IA infusion). Then, IV nicotine will be administered (0.5-1.5 mg/70 kg will be infused over 10 minutes). Following a series of 4 nicotine vaccine shots, the same procedure will be repeated for a second [123I]5-IA scan day. We hypothesize that occupancy of β2-nAChR will be significantly lower, and take longer to plateau, following nicotine vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker who smokes at least 10-25 cigarettes a day
* Good general health

Exclusion Criteria:

* Subjects with a pacemaker or other ferromagnetic material in body.
* Prior exposure to NicVAX or any other nicotine vaccine.
* Use of systemic steroids or other immunosuppressive agent
* History of significant neurological, cardiovascular, hepatic, endocrine, renal, liver, psychiatric or thyroid illness
* Cancer or cancer treatment in last 5 years
* HIV infection
* Use of varenicline (Chantix), bupropion (Wellbutrin, Zyban), mecamylamine (Inversin), within 30 days prior to administration of NicVAX and for the duration of the study.
* Inability to fulfill all visits and examination procedures for approximately 20 weeks.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irina Esterlis, Ph.D., Principal Investigator — Yale University
Locations (1):
- Veterans Association Connecticut Hospital System, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Esterlis I, Hannestad JO, Perkins E, Bois F, D'Souza DC, Tyndale RF, Seibyl JP, Hatsukami DM, Cosgrove KP, O'Malley SS. Effect of a nicotine vaccine on nicotine binding to beta2*-nicotinic acetylcholine receptors in vivo in human tobacco smokers. Am J Psychiatry. 2013 Apr;170(4):399-407. doi: 10.1176/appi.ajp.2012.12060793. PMID 23429725

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment in to the study ended in Feb. 2011. Subjects were screened and recruited from the VA West Haven, CT.
Pre-assignment Details: Several possible subject were not enrolled in to the study because of the exclusion/inclusion criteria, such as allergies to medications, high blood pressure, or SCID II diagnosis
Groups:
- Healthy Smoker: Healthy smokers with nicotine dependence
  Nicotine bitartrate : 0.5-1.5 mg of Nicotine bitartrate, I.V. on each of two SPECT Scan days
  [123I]5-IA-85380 : up to 10 mCi of [123I]5-IA-85380, I.V. on each of two SPECT Scan days
  NicVAX : 1.0 mL of Nicotine Conjugate Vaccine(x4), I.M. at 3 week intervals between SPECT studies
Period: Overall Study
Arm/Group | Healthy Smoker
Started | 14
Completed | 11
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — withdrawn by PI | 1

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Smoker
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.15 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Mean of the Average Nicotine Binding % at Scan 1 and Scan 2
Description: nAchR levels from baseline and after immunization with 3'-AmNic-rEPA (NicVAX=vaccine) SPECT images obtained in healthy control smoking subjects at baseline and after immunization with 3'-AmNic-rEPA (NicVAX=vaccine). nAchR levels will be determined by radioligand uptake in SPECT images. Means were calculated for all subjects at scan 1 and scan 2.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of average nicotine binding
Arm/Group | Healthy Smoker
Number analyzed (Participants) | 11
percentage of average nicotine binding
  Scan 1 | 54.9 (8.7)
  Scan 2 | 49.1 (10.1)
Statistical Analysis 1: Comparison: Healthy Smoker; This is a comparison of scan 1 and scan 2; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | Healthy Smoker
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor has 30 days to approve anything that PI would like to publish and/or present